CLINICAL TRIAL: NCT03360942
Title: Long Term Follow-up of Deep Brain Stimulation for Treatment-Resistant Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D12131; 23442 (Other: Dartmouth Committee for the Protection of Human Subjects)
Record Dates: First submitted 2017-08-17; First posted 2017-12-04 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-08

CONDITIONS: Treatment Resistant Depression; Depressive Disorder, Treatment-Resistant; Depression, Bipolar
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DBS Long Term Follow Up (Experimental): 5 participants who were in a prior study to receive DBS are enrolled to have their progress and DBS devices monitored for a period of 12 years.
  Interventions: Device: SCC DBS

INTERVENTIONS:
Device: SCC DBS — Deep Brain Stimulator
  Other Names: Libra(TM) Implantable Deep Brain Stimulation (DBS) System

SUMMARY:
The long term follow up of a pilot study in which the investigators proposed to test whether high frequency stimulation of the subcallosal cingulate (SCC) is a safe and efficacious antidepressant treatment in five TRD patients, to compare the effects of left-sided vs. right-sided stimulation, and to investigate potential mechanisms of action of this intervention. Importantly, this study will be used to assess the need for and assist in planning a larger, more definitive trial of SCC Deep Brain Stimulation (DBS) for treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
The U.S. lifetime prevalence of major depressive disorder (MDD) is 17%. A number of treatments are available for depression including medications, psychotherapy and various somatic treatments. Unfortunately, up to two-thirds of patients remain symptomatic following first-line treatment and a third fail to achieve remission (defined as full resolution of depressive symptoms) after four established treatments; approximately 10%-20% of depressed patients may show virtually no improvement despite multiple, often aggressive treatments. Thus, a conservative estimate places the U.S. prevalence of treatment-resistant depression (TRD) at 1%-3%. TRD has a high risk of suicide, is a major cause of disability and is responsible for doubling of overall health care costs.

For patients with TRD there are limited evidence-based treatment options. Transcranial magnetic stimulation (TMS) may have efficacy for patients that have failed no more than one antidepressant medication 10-12, but response and remission rates are relatively low (under 30% and 20% respectively). Vagus nerve stimulation (VNS) may have efficacy in patients that have failed 4-6 antidepressant treatments but long-term response and remission rates are again low (about 20% and 10% respectively). Electroconvulsive therapy(ECT) can be effective in TRD patients with remission rates of 50%-60%. However, more than 70% of TRD patients will relapse within 6 months following a successful acute treatment course. For patients that have failed ECT, there are no evidence-based treatment options. Therefore, there is great need for novel treatment approaches for TRD.

Prior clinical trials have shown that SCC DBS has the potential to be a valuable treatment option for patients with TRD. Further developing this treatment will involve confirming its effectiveness and identifying ways to optimize its use. In this study the investigators intend to test the safety and efficacy of chronic SCC DBS as a treatment for TRD and compare the safety and efficacy of left-sided versus right-sided stimulation using a double-blind, randomized, cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Have received DBS for TRD
* Ability to provide written informed consent
* Willing to comply with all necessary study visits

Exclusion Criteria:

* Significant cerebrovascular risk factors or a previous stroke, documented major head trauma or neurodegenerative disorder.
* Other currently active clinically significant Axis I psychiatric diagnosis including schizophrenia, panic disorder, obsessive-compulsive disorder, generalized anxiety disorder or post-traumatic stress disorder. Patients with severe Axis II personality disorders will also be excluded if the personality disorder is likely to interfere with cooperation and adherence to the study protocol.
* Current psychotic symptoms.
* Evidence of global cognitive impairment.
* Substance abuse or dependence not in full sustained remission (i.e., not active for at least one year).
* Active suicidal ideation with intent; suicide attempt within the last six months; more than three suicide attempts within the last two years.
* Pregnancy or plan to become pregnant during the study period.
* General contraindications for DBS surgery (cardiac pacemaker/defibrillator or other implanted devices).
* Inability or unwillingness to comply with long-term follow-up.
* History of intolerance to neural stimulation of any area of the body.
* Participation in another drug, device or biologics trial within the preceding 30 days.
* Conditions requiring repeated MRI scans.
* Conditions requiring diathermy.
* Conditions requiring anticoagulant medication.
* Terminal illness associated with expected survival of <12 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 participants were in a prior study (NCT01898429) to receive Deep Brain Stimulation (DBS) and were asked to enroll to have their progress and DBS devices monitored for a period of 12 years.
Groups:
- DBS Long Term Follow Up: Participants with Deep Brain Stimulation for Treatment-Resistant Depression
Period: Overall Study
Arm/Group | DBS Long Term Follow Up
Started | 5
Completed | 0
Not Completed | 5
Not completed — Device explanted | 2
Not completed — Study closure | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Device Was Functioning
Description: Patients will be evaluated every 12 months by the study psychiatrist (via in-person, phone or video call visit) to assess device functioning,
Time Frame: Data was to be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months); Data were collected from 1 to 6 years.
Population: One participant had the device explanted after one year of follow-up, and thus the number analyzed dropped from 5 to 4 after the first year. After the 5th year assessment, one additional participant had the device explanted, and one participant withdrew from participation dropping the number of participants analyzed from 4 to 2. The study was closed after the sixth year.
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 5
Participants
  Year 1: Yes Functioning | 3
  Year 1: No, Not Functioning | 1
  Year 1: Unknown (No data recorded regarding status of device) | 1
  Year 2: number analyzed (Participants) | 4
  Year 2: Yes Functioning | 2
  Year 2: No, Not Functioning | 0
  Year 2: Unknown (No data recorded regarding status of device) | 2
  Year 3: number analyzed (Participants) | 4
  Year 3: Yes Functioning | 1
  Year 3: No, Not Functioning | 0
  Year 3: Unknown (No data recorded regarding status of device) | 3
  Year 4: number analyzed (Participants) | 4
  Year 4: Yes Functioning | 1
  Year 4: No, Not Functioning | 0
  Year 4: Unknown (No data recorded regarding status of device) | 3
  Year 5: number analyzed (Participants) | 4
  Year 5: Yes Functioning | 1
  Year 5: No, Not Functioning | 0
  Year 5: Unknown (No data recorded regarding status of device) | 3
  Year 6: number analyzed (Participants) | 2
  Year 6: Yes Functioning | 0
  Year 6: No, Not Functioning | 0
  Year 6: Unknown (No data recorded regarding status of device) | 2

2. Primary Outcome: Mean Hamilton Depression Rating Scale (HDRS-17) Score Over Time
Description: The Hamilton Depression Rating Scale-17 (HDRS-17) is a 17-item clinician-administered depression assessment scale pertaining to symptoms of depression experienced over the past week. For the HDRS-17, a score of 0-7 is generally accepted to be within the normal range., a score of 8-12: Possible depression, a score of 13-17: Mild depression, a score of 18-24: Moderate depression, a score of 25-52: Severe depression.
Time Frame: Data was to be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months); Data were collected for 1 to 2 years.
Population: In year 1, confirmation of psychiatrist oversight or completion of assessment could not be verified for 3 of 5 participants. One participant had device explanted after year 1 and no data was collected for this participant thereafter. Data for 2 of 4 participants were not collected utilizing this tool after year 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants for year 2. No data was collected utilizing this assessment after year 2.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
score on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 18 [16 to 20]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 24 [24 to 24]

3. Primary Outcome: Mean Hamilton Depression Rating Scale-21 (HDRS-21) Score Over Time
Description: The Hamilton Rating Scale for Depression or Hamilton Depression Rating scale (HDRS-21) is a 21-item clinician-administered multiple-choice measure of depression symptom severity. The scale consists of 21 items assessing various aspects of depression, including mood, guilt, insomnia, agitation & anxiety. Participants are rated on each item based on the presence & severity of symptoms, with scores ranging from 0 to 2 or 0 to 4. The first 17 items measure the severity of depressive symptoms & the scores from those 17 items are combined to create a total score (52 max). Higher total scores indicate more severe depression, with ranges typically interpreted as follows: a score of 0-7 is generally accepted to be within the normal range (Minimal or no depression), a score of 8-13: Mild depression, a score of 14-18: Moderate depression, a score of 19-22: Severe depression, a score of 23 and above: very severe depression. The sum of all 21 items results in highest possible score of 76.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
units on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 22 [20 to 24]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 25 [25 to 25]

4. Primary Outcome: Mean Hamilton Depression Rating Scale-24 (HDRS-24) Score Over Time
Description: The Hamilton Rating Scale for Depression or Hamilton Depression Rating scale (HDRS-24) is a 24-item clinician-administered multiple-choice measure of depression symptom severity. The scale consists of 24 items that assess various aspects of depression, including mood, guilt, insomnia, agitation, and anxiety. Participants are rated on each item based on the presence and severity of symptoms, with scores ranging from 0 to 2 or 0 to 4. The first 17 items measure the severity of depressive symptoms, and the scores from those 17 items are combined to create a total score (52 max). Higher total scores on the HDRS-24 indicate more severe depression, with ranges typically interpreted as follows: 0-7 (normal), 8-13 (mild depression), 14-18 (moderate depression), 19-22 (sever depression) and 23 or higher (very severe depression). The sum of the scores from all 24 items results in the highest possible score being 78.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
score on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 29.5 [27 to 32]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 28 [28 to 28]

5. Primary Outcome: Mean Hamilton Depression Rating Scale-28 (HDRS-28) Score Over Time
Description: The Hamilton Rating Scale for Depression or Hamilton Depression Rating scale (HDRS-28) is a 28-item clinician-administered multiple-choice measure of depression symptom severity. The scale consists of 28 items that assess various aspects of depression, including mood, guilt, insomnia, agitation, and anxiety. Participants are rated on each item based on the presence and severity of symptoms, with scores ranging from 0 to 2 or 0 to 4. The first 17 items measure the severity of depressive symptoms, and the scores from those 17 items are combined to create a total score (52 max). Higher total scores on the HDRS-28 indicate more severe depression, with ranges typically interpreted as follows: 0-7 (normal), 8-13 (mild depression), 14-18 (moderate depression), 19-22 (Sever depression) and 23 or higher (very severe depression). The sum of the scores from all 28 items results in the total score, with the highest possible score being 84.
Time Frame: Data was to be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months); Data were collected at 1 year after impanation or 2 years after implantation.
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
score on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 32.5 [30 to 35]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 31 [31 to 31]

6. Primary Outcome: Mean Montgomery-Åsberg Depression Rating Scale (MADRS) Score Over Time
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinical assessment tool used to measure the severity of depressive symptoms in individuals diagnosed with depression. The scale consists of 10 items that assess various symptoms of depression, including apparent sadness, reported sadness, inner tension, sleep disturbances, and reduced appetite. Each item is rated on a scale from 0 to 6, with higher scores indicating more severe symptoms. The total score on the MADRS ranges from 0 to 60, with higher scores reflecting greater severity of depression. Interpretation of MADRS scores is as follows: 0-6 (normal), 7-19 (mild depression), 20-34 (moderate depression), and 35 or higher (severe depression).
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
score on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 25 [24 to 26]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 25 [25 to 25]

7. Primary Outcome: Mean Hamilton Anxiety Rating Scale Over Time
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items, each of which assesses a different symptom of anxiety. These items cover both psychological and physical manifestations of anxiety. Each item is scored on a scale from 0 to 4, with 0 indicating the absence of the symptom and 4 indicating severe or disabling symptoms. The total score can range from 0 to 56, with higher scores indicating more severe anxiety.
Time Frame: as for outcome 5
Population: 1 of 5 participants did not have this data collected at any time. In year 1, confirmation of psychiatrist oversight/completion of assessment could not be verified for 3 of 4 participants. After year 1, data for 2 participants were not collected. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants for year 2. No data was collected after year 2.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
units on a scale
  Year 1: number analyzed (Participants) | 1
  Year 1 | 25 [25 to 25]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 25 [25 to 25]

8. Primary Outcome: Mean Young Mania Rating Scale (YMRS) Score Over Time
Description: The Young Mania Rating Scale (YMRS) is a clinical assessment tool designed to measure the severity of manic symptoms in individuals diagnosed with bipolar disorder. The scale consists of an 11-item scale used to assess the severity of manic states, including elevated mood, increased energy levels, irritability, impulsivity, and grandiosity. Four items are graded on a scale of 0 to 8 (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a scale of 0 to 4. Higher scores indicating more severe manic symptoms. The total score on the YMRS ranges from 0 to 60, with higher scores reflecting greater severity of mania. Interpretation of YMRS scores is as follows: 0-12 (normal), 13-20 (mild mania), 21-35 (moderate mania), and 36 or higher (severe mania).
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
score on a scale
  Year 1: number analyzed (Participants) | 1
  Year 1 | 0 [0 to 0]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 0 [0 to 0]

9. Primary Outcome: Mean Beck Depression Inventory-II (BDI-II) Score Over Time
Description: The Beck Depression Inventory-II (BDI-II) is a self-report questionnaire designed to assess the severity of depressive symptoms in individuals aged 13 and older. The scale consists of 21 items that measure various symptoms of depression, such as mood, pessimism, guilt, and physical symptoms. Participants rate each item based on how they have been feeling over the past two weeks, with scores ranging from 0 to 3. Higher total scores on the BDI-II indicate more severe depressive symptoms, with ranges typically interpreted as follows: 0-13 (minimal depression), 14-19 (mild depression), 20-28 (moderate depression), and 29-63 (severe depression).
Time Frame: Data was to be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months). Data were collected at 1 year after impanation or 2 years after implantation.
Population: as for outcome 7
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
score on a scale
  Year 1: number analyzed (Participants) | 1
  Year 1 | 36 [36 to 36]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 26 [26 to 26]

10. Primary Outcome: Mean Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) Score Over Time
Description: The Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) is a clinical assessment tool used to measure the severity of depressive symptoms in individuals diagnosed with depression. The scale consists of 16 items that assess nine criterion symptom domains of depression according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria. Participants rate each item based on how they have been feeling over the past seven days, with scores ranging from 0 to 3 or 0 to 4. Higher total scores on the QIDS-SR indicate more severe depressive symptoms, with ranges typically interpreted as follows: 0-5 (no depression), 6-10 (mild depression), 11-15 (moderate depression), 16-20 (severe depression), and 21-27 (very severe depression).
Time Frame: Data will be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months); Data were collected at 1 year after impanation or year 2 and 3 after implantation.
Population: In year 1 confirmation of psychiatrist oversight/completion of assessment could not be verified for 3 of 5 participants. 1 participant had device explanted after year 1 & no data was collected thereafter. Data for 2 of 4 participants were not collected utilizing this tool after yr 1. In year 2 confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants. Data for 1 of 2 participants were not collected after yr 2. No data was collected after yr 3.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
units on a scale
  Year 1: number analyzed (Participants) | 2
  Year 1 | 16 [16 to 16]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 15 [15 to 15]
  Year 3: number analyzed (Participants) | 1
  Year 3 | 9 [9 to 9]

11. Primary Outcome: Mean Global Assessment of Functioning (GAF) Score Over Time
Description: The Global Assessment of Functioning (GAF) is a single-item mental health status measure which assesses how much a person's symptoms affect their day-to-day life on a scale of 0 to 100. Higher scores indicating better overall functioning.
Time Frame: Data will be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months); Data were collected at 1 year after impanation or 2 years after implantation.
Population: 3 of 5 participants enrolled in this study did not have this data collected at any time. In year 1, confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants. Data for one participant was not collected utilizing this assessment tool after year 1. No data was collected after the second year for the entire cohort utilizing this assessment tool.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
units on a scale
  Year 1: number analyzed (Participants) | 1
  Year 1 | 55 [55 to 55]
  Year 2: number analyzed (Participants) | 1
  Year 2 | 65 [65 to 65]

12. Primary Outcome: Number of Participants Reporting Suicidal Behavior or Actual Attempts Using the Columbia- Suicide Severity Rating Scale (C-SSRS) Over Time
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinical assessment tool used to evaluate the severity of suicidal ideation and behavior in individuals. The scale consists of several items that assess suicidal ideation, suicidal behavior, and the severity of suicidal intent. Scores on the C-SSRS are not summed to provide a total score; instead, each item is scored individually to assess presence, frequency, and severity of suicidal thoughts or actions.
Time Frame: Data will be collected every year (approximately every 12 months) for up to 10 Years after the implantation of the device (approximately 120 months). Data were collected at 1 year after impanation or 2 years after implantation.
Population: 1 of 5 participants did not have this data collected at any time. 1 of 4 participants did not have this data collected in yr 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 3 participants in yr 1. 1 participant had device explanted and data for 1 of 3 participants were not collected after yr 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants for yr 2. No data was collected after yr 2.
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 3
Participants
  Year 1: number analyzed (Participants) | 2
  Year 1 | 0
  Year 2: number analyzed (Participants) | 1
  Year 2 | 0

13. Primary Outcome: Number of Participants Reporting a Specific Value in the Severity of Illness Section of the Clinical Global Impressions (CGI) Assessment
Description: The Clinical Global Impression (CGI) is a standardized assessment tool used to provide a global evaluation of illness severity and treatment response in individuals with mental health disorders. The CGI consists of two main scales: the Clinical Global Impression-Severity (CGI-S) scale and the Clinical Global Impression-Improvement (CGI-I) scale. CGI-Scale: The CGI-S scale is used to assess the severity of illness at a specific point in time. The range of responses for the Severity of Illness section of the CGI are: Normal, not at all ill, Borderline mentally ill, Mildly ill, Moderately ill, Markedly ill, Severely ill, Among the most extremely ill patients. This outcome measure reports the number of participants for whom data was available and the specific response for this section of the CGI.
Time Frame: as for outcome 12
Population: 2 of 5 participants did not have this data collected at any time. 1 of 3 participants did not have this data collected in year 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants in year 1. Data for 1 of 3 participants were not collected after year 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants for year 2. No data was collected after year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
Participants
  Year 1: number analyzed (Participants) | 1
  Year 1: Moderately Ill | 1
  Year 1: Mildly Ill | 0
  Year 2: number analyzed (Participants) | 1
  Year 2: Moderately Ill | 0
  Year 2: Mildly Ill | 1

14. Primary Outcome: Number of Participants Reporting a Specific Value in the Global Improvement Section of the Clinical Global Impressions Assessment
Description: The Clinical Global Impression (CGI) is a standardized assessment tool used to provide a global evaluation of illness severity and treatment response in individuals with mental health disorders. The CGI consists of two main scales: the Clinical Global Impression-Severity (CGI-S) scale and the Clinical Global Impression-Improvement (CGI-I) scale. CGI-Scale: The CGI-I scale is used to assess the overall improvement or change in symptoms over time in response to treatment. The range of responses for the CGI-I are: Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse. This outcome measure reports the number of participants for whom data was available and the specific response for this section of the CGI.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
Participants
  Year 1: number analyzed (Participants) | 1
  Year 1: Much improved | 0
  Year 1: Minimally improved | 1
  Year 2: number analyzed (Participants) | 1
  Year 2: Much improved | 1
  Year 2: Minimally improved | 0

15. Primary Outcome: Number of Participants Providing a Specific Response Using the Patient Global Impressions (PGI) of Change Scale
Description: The Patient Global Impression (PGI) is a self-reported assessment tool used to measure the overall severity of illness or improvement in symptoms from the patient's perspective. The potential responses to the PGI are Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, Very Much Worse. This outcome measure reports the number of participants for whom data was available.
Time Frame: as for outcome 12
Population: 2 of 5 participants did not have this data collected at any time. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 2 of 3 participants in year 1. Data for 1 of 3 participants were not collected after year 1. Confirmation of psychiatrist oversight/completion of assessment could not be verified for 1 of 2 participants for year 2. No data was collected after year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
Participants
  Year 1: number analyzed (Participants) | 1
  Year 1: Much Improved | 1
  Year 1: Minimally Improved | 0
  Year 2: number analyzed (Participants) | 1
  Year 2: Much Improved | 0
  Year 2: Minimally Improved | 1

16. Primary Outcome: Number of Participants Providing a Specific Response Using the Patient Global Impressions (PGI) of Severity Scale
Description: The potential responses to the Patient Global Impressions of Severity scale are Normal, not at all ill, Borderline mentally ill , Mildly ill, Moderately ill, Markedly ill, Severely ill, Among the most extremely ill patients. This outcome measure reports the number of participants for whom data was available and the specific response for this section of the PGI
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | DBS Long Term Follow Up
Number analyzed (Participants) | 2
Participants
  Year 1: number analyzed (Participants) | 1
  Year 1: Mildly Ill | 1
  Year 1: Markedly Ill | 0
  Year 2: number analyzed (Participants) | 1
  Year 2: Mildly Ill | 0
  Year 2: Markedly Ill | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment up to two years, on average. One participant had the device explanted after one year, and no adverse events were collected for this participant after the first year.
Groups:
- DBS Long Term Follow Up: 5 participants who were in a prior study to receive DBS are enrolled to have their progress and DBS devices monitored for a period of 12 years.
  DBS: Deep Brain Stimulator
Arm/Group | DBS Long Term Follow Up
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS Long Term Follow Up (N=5)
Hospitalization (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS Long Term Follow Up (N=5)
Trouble Sleeping (Psychiatric disorders) | 4 (6)
Nightmares or other sleep disturbance (Psychiatric disorders) | 3 (4)
Feeling drowsy or sleepy (Nervous system disorders) | 3 (4)
Feeling nervous or hyper (Psychiatric disorders) | 4 (4)
Weakness or fatigue (Musculoskeletal and connective tissue disorders) | 3 (4)
Irritable (Psychiatric disorders) | 3 (4)
Poor memory (Nervous system disorders) | 3 (4)
Trouble concentrating (Nervous system disorders) | 2 (4)
Feeling strange (Psychiatric disorders) | 2 (2)
Numbness or tingling (Nervous system disorders) | 3 (3)
Dizziness or faintness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (7)
Blurred vision (Eye disorders) | 2 (2)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 4 (5)
Drooling or increased salivation (Nervous system disorders) | 1 (1)
Muscle cramps or stiffness (Musculoskeletal and connective tissue disorders) | 2 (3)
Trouble sitting still (Psychiatric disorders) | 3 (4)
Tremor or shakiness (Nervous system disorders) | 2 (3)
Poor coordination or unsteadiness (Nervous system disorders) | 2 (3)
Heartbeat rapid or pounding (Cardiac disorders) | 3 (4)
Trouble catching breath or hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nausea or vomiting (Gastrointestinal disorders) | 2 (3)
Stomach or abdominal discomfort (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Frequent need to urinate (Renal and urinary disorders) | 2 (2)
Loss of sexual interest (Psychiatric disorders) | 2 (3)
Problems with sexual arousal (erection or lubrication) (Psychiatric disorders) | 3 (4)
Delayed or absent orgasm (Psychiatric disorders) | 3 (4)
Sweating excessively (Skin and subcutaneous tissue disorders) | 2 (3)
Fluid retention or swelling (General disorders) | 3 (3)
Appetite decreased (Metabolism and nutrition disorders) | 1 (2)
Appetite increased (Metabolism and nutrition disorders) | 2 (2)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (2)
Skin rash or allergy (Immune system disorders) | 3 (4)
Diminished mental acuity/sharpness (Nervous system disorders) | 2 (3)
Difficulties finding words (Nervous system disorders) | 3 (4)
Apathy/Emotional Indifference (Psychiatric disorders) | 2 (3)
Dizziness when you stand up (Nervous system disorders) | 3 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Hair thinning/loss (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (2)
Clenching of teeth at night (Psychiatric disorders) | 4 (5)
Strange taste in mouth (Nervous system disorders) | 1 (2)
Unable to sit still (Psychiatric disorders) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Felt Sick (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03360942/Prot_SAP_000.pdf